CLINICAL TRIAL: NCT03281408
Title: Perioperative Obstructive Sleep Apnea Intervention Study
Brief Title: Perioperative Complications and Myocardial Injury Risk in Arthoplasty Patients Suspected of Having Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other)
Responsible Party: Principal Investigator, Steven Lee, Clinical Assistant Professor, University of British Columbia
Other Study IDs: H17-01022
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Suspected OSA Patients Undergoing Knee or Hip Arthroplasty: These 100 subjects will be cared for and monitored in hospital following current hospital protocol. No change or intervention is to be administered. Troponin testing will be done post-op with other routine blood work.

SUMMARY:
Obstructive Sleep Apnea (OSA) is a common and under-diagnosed breathing disorder characterized by recurrent partial or complete collapse of the upper airway (tongue, soft palate) during sleep. It causes recurrent episodes of asphyxia (suffocation) resulting in fragmented sleep, low blood oxygen levels (hypoxemia), and high carbon dioxide concentrations. Untreated OSA is associated with serious heart/lung and metabolic diseases including strokes, diabetes, and heart attacks.

When a patient with OSA undergoes surgery, the symptoms of OSA are exacerbated afterwards due to the effects of anesthesia and related medications such as those used for pain control. This puts patients at higher risk for complications and necessitates nursing care and monitoring that are resource intensive. In many hospitals, patients with an OSA diagnosis are monitored after surgery in "high acuity" wards where the nurse to patient ratio is higher than usual. These high acuity/monitored beds are often in high demand, and their unavailability may sometimes mean cancellation of surgery or prolonged patient stay in the Post-operative Recovery Room, further causing operating room backlog.

Another serious issue is that many patients do not know they actually have the OSA condition. It is estimated that up to 20% (1) of people in the general public have OSA and that 75% (2) of them are not diagnosed. When someone with OSA goes for surgery without previously being diagnosed, special precautions in care and monitoring may not be in place, until a complication develops. For this reason, this population - those most susceptible to have OSA, but with no previous formal testing for the condition - is the most at risk for complications, and is the target group for this trial.

We plan to identify the study population by screening for OSA using the STOP-BANG questionnaire. Those who score high on this 8 item screening test have high likelihood of actually having OSA if they were to undergo formal testing and diagnosis in a Sleep Lab.

We will identify cardio-respiratory complications by conducting a chart review and determine whether admission to a "high acuity" bed had any impact. As OSA patients are at higher risk for cardiovascular complications at baseline and around the time of surgery, blood test for troponin will be performed on post-op day 1 and 2 to investigate the rate of myocardial injury. With the rate of MINS (myocardial injury after non-cardiac surgery) reported to be 8% with almost 10% 30 day mortality (per VISION trial), this pilot project which focuses on arthroplasty patients with suspected OSA, will inform us of the arthroplasty surgery specific MINS risk for comparison.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective primary or revision knee/hip replacement surgery.
2. Patients with no previous OSA diagnosis (by polysomnography), who score >=5 on STOP-BANG OSA screening.

Exclusion Criteria:

1. Patients without ability to communicate in English by reading or writing.
2. Patients with renal failure.
3. Patients on CPAP therapy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the UBC Hospital to have knee/hip arthroplasty surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Composite Adverse Events | 0-96 hours
  The incidence of adverse events (each listed as a secondary outcome) related to OSA combined as a composite end point
Troponin | Post-op Day 1
  Testing for risk of MINS (myocardial injury after non-cardiac surgery)
Troponin | Post-op Day 2
  Testing for risk of MINS (myocardial injury after non-cardiac surgery)

SECONDARY OUTCOMES:
Respiratory or Cardiac Arrest | 0-96 hours
  Activation of Code Blue
Respiratory Therapy beyond standard nasal prong oxygen | 0-96 hours
Pneumonia | 0-96 hours
  Fever with temp >=38 degree Celsius, leukocytosis and new infiltrate on CXR
Naloxone Usage | 0-96 hours
  For opioid reversal
Airway Intervention for any cause | 0-96 hours
  Use of nasal/oral airway or intubation, jaw thrust/chin lift
Cardiac Arrhythmia | 0-96 hours
  New arrhythmia requiring treatment
Cardiac ischemia or injury | 0-48 hours
  ECG changes or troponin elevation
Transfer from normal ward bed to monitored bed | 0-96 hours
Transfer to local tertiary hospital | 0-96 hours

OTHER OUTCOMES:
30 Day Mortality | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- UBC Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peppard PE, Young T, Barnet JH, Palta M, Hagen EW, Hla KM. Increased prevalence of sleep-disordered breathing in adults. Am J Epidemiol. 2013 May 1;177(9):1006-14. doi: 10.1093/aje/kws342. Epub 2013 Apr 14. PMID 23589584
- [Background] Punjabi NM. The epidemiology of adult obstructive sleep apnea. Proc Am Thorac Soc. 2008 Feb 15;5(2):136-43. doi: 10.1513/pats.200709-155MG. PMID 18250205